CLINICAL TRIAL: NCT00664820
Title: Effects of Probiotics on Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); St. Joseph's Health Care London (Other)
Responsible Party: Principal Investigator, Gregor Reid, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R-08-140
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritics; probiotics; Lactobacillus
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Will receive two Urex-CAP-5 (probiotic Lactobacillus rhamnosus GR-1 and L. reuteri RC-14) capsules daily for 3 months.
  Interventions: Dietary Supplement: Probiotic capsules containing Lactobacillus rhamnosus GR-1 and L. reuteri RC-14

INTERVENTIONS:
Dietary Supplement: Probiotic capsules containing Lactobacillus rhamnosus GR-1 and L. reuteri RC-14 — 2 capsules daily for 3 months.
  Other Names: Urex-CAP-5 capsule

SUMMARY:
The purpose of the present study is to examine the utility of probiotics as an adjunctive therapy (in addition to patients' pharmacotherapy) for the treatment of Rheumatoid Arthritis.

We hypothesize that specifically selected probiotics, Lactobacillus rhamnosus GR-1 and L. reuteri RC-14, can alleviate symptoms of RA and thereby increase the daily activity of these patients.

DETAILED DESCRIPTION:
Patients between 18 - 80 years old who have Rheumatoid arthritis with at least 4 swollen and tender joints will be randomized to receive by mouth two capsules containing placebo or probiotic, Lactobacillus rhamnosus GR-1 and L. reuteri RC-14, daily. The subjects will continue to take the placebo or probiotic, in addition to their RA medications (i.e. ongoing medication and/or other therapy, such as physiotherapy are permitted, except immunotherapy) for three months.

At day 0 (visit #1) (when recruited and just prior to starting to take capsules), at day 45 (visit #2), and at day 90 (visit #3), blood samples of approximately 40 ml of blood (8 teaspoons) will be collected by clinical technicians working in the Lab Test Centre at St. Joseph's Health Center. The blood samples will be used to evaluate Erythrocyte Sedimentation Rate (ESR) and C-reactive protein level. In addition, immunological markers like TNFα, IL-12, IL-10 and G-CSF will also be measured. Serum creatinine and liver function will be evaluated as parameters of any side effects of the probiotics.

Probiotics/placebo will be dispensed from the pharmacy and provided to the subjects by the study investigator at the first visit (for the first 45 days) and second visit (for the final 45 days).

At day 0, 45 and 90 (visits 1, 2 and 3) a physical exam will be completed, where the physician will count the number of swollen and tender joints and complete the Physician Global Assessment of Disease activity. In addition, at these times, the patients will be asked to complete the following self-administered questionnaires:

* Health Assessment Questionnaire (HAQ);
* Patient's Global Assessment of Disease Activity
* Patient Assessment of Pain and Assessment of Duration of Morning stiffness.

Patients will also be asked about feeling fatigued or sleepy, as these are standard questions that come with the above-mentioned questionnaires. These are simple questionnaires that will take approximately 15 minutes to complete. In visit 2 and 3 the physician will confirm if the participant is taking the study capsule/placebo correctly, review any new medications the patient has taken since the last visit and will ask about adverse events that may have occurred.

At day 90, subjects will stop taking capsules.

A follow-up phone call will take place 30 days after the completion of the study medication (day 120). If a patient is withdrawn or withdraws from the study prematurely, he/she will be asked to receive a follow-up telephone call 30 days from the date they last took the study product. During the phone call, which should not take more than 10 minutes, the participant will be asked about any medications taken in the past month and about any possible side effects (unwanted effects or health problems) that they may have experienced.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the ages of 18 to 80
2. Are clinically diagnosed with RA (according to ACR criteria)
3. Have been on stable RA treatment and are expected to stay on stable RA treatment during the time of the study (i.e. ongoing medication and/or other therapy, such as physiotherapy are permitted, except immunotherapy).
4. Have at least 4 swollen and tender joints on a 64/66 scale
5. Women of childbearing capacity and who agree to an acceptable method of birth control. Acceptable methods of birth control will include: hormone therapy (oral birth control pills, injectable or skin patches), barrier contraceptive with spermacide, an intra uterine device (IUD) or complete abstinence (no sexual intercourse).
6. Patients who did not meet any of the exclusion criteria stated below.

Exclusion Criteria:

1. Receiving ongoing immunotherapy for RA
2. Has inflammatory bowel disease or leaky gut
3. Currently consuming probiotics and refuse to have a two week washout period
4. Have known allergies to any component in the study product or placebo
5. Plan to have surgery during the time of the study
6. Mental illness impairing ability to comply with study
7. Women who are pregnant or plan to get pregnant during the study period
8. Women who are breastfeeding
9. Consumption of probiotic-containing products during study treatment
10. Patients participating in another NHP clinical trial
11. Patients enrolled in another clinical trial in the past 3 month
12. Women who are breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the number of patients that achieve an ACR20 response. So we will compare the number of patients that achieved an ACR20 response in the probiotic group to those that achieved an ACR20 response in the placebo group. | 4 months

SECONDARY OUTCOMES:
Immunological parameters (TNFα, IL-12, IL-10 and G-CSF) along with the eight components of the ACR20 response will be the secondary outcomes. Serum creatinine and liver function will be evaluated as parameters of any side effects of the probiotics. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pineda, BA, Study Director — Western University, Canada; Janet Pope, MD, Study Director — St. Joseph's Health Center; Gregor Reid, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada